CLINICAL TRIAL: NCT02336594
Title: A Phase 1, Randomized, Open-Label, Crossover Study in Healthy Adult Male Subjects to Assess the Relative Bioavailability of Two RDEA3170 Tablets
Brief Title: RDEA3170 Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA3170-110
Record Dates: First submitted 2014-11-06; First posted 2015-01-13 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence ABCD (Experimental): 2.5 mg x 4 tablets qd (once daily) fasted, 10 mg tablet qd fasted, 10 mg tablet qd fed low-fat, 10 mg tablet qd fed high-fat.
  Interventions: Drug: RDEA3170 10 mg; Drug: RDEA3170 2.5 mg
- Sequence BACD (Experimental): 10 mg tablet qd fasted, 2.5 mg x 4 tablets qd fasted, 10 mg tablet qd fed low-fat, 10 mg tablet qd fed high-fat
  Interventions: Drug: RDEA3170 10 mg; Drug: RDEA3170 2.5 mg
- Sequence ABDC (Experimental): 2.5 x 4 mg tablets qd fasted, 10 mg tablet qd fasted, 10 mg tablet qd fed high-fat, 10 mg tablet qd fed low-fat
  Interventions: Drug: RDEA3170 10 mg; Drug: RDEA3170 2.5 mg
- Sequence BADC (Experimental): 10 mg tablet qd fasted, 2.5 mg x 4 tablets qd fasted, 10 mg tablet qd fed high-fat, 10 mg tablet qd fed low-fat
  Interventions: Drug: RDEA3170 10 mg; Drug: RDEA3170 2.5 mg

INTERVENTIONS:
Drug: RDEA3170 10 mg
Drug: RDEA3170 2.5 mg

SUMMARY:
This is a Phase 1, randomized, open-label, 4-way crossover pharmacokinetic (PK) and pharmacodynamic (PD) study in healthy adult male subjects designed to assess the relative bioavailability of RDEA3170 2.5 mg tablets administered as a 10 mg dose (2.5 mg × 4 tablets) and of a single RDEA3170 10 mg tablet. This study will also assess the effect of a low-fat and high-fat meal on the PK and PD of RDEA3170 10 mg tablets.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures and the risks involved and is willing to provide written informed consent before the first study-related activity
* Subject has a body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 40 kg/m2
* Subject has a Screening serum urate level ≤ 7 mg/dL
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment

Exclusion Criteria:

* Subject has a history or suspicion of kidney stones
* Subject has undergone major surgery within 3 months prior to Screening
* Subject donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to Day 1
* Subject has inadequate venous access or unsuitable veins for repeated venipuncture
* Subject has a Screening serum creatinine value above the upper limit of normal during Screening or at Day -2 (Admission)
* Subject cannot swallow multiple tablets
* Subject is a heavy caffeine drinker
* Subject is unwilling to comply with the dietary restrictions of the study
* Subject is unable or unwilling to comply with the study requirements or has a situation or condition that, in the opinion of the Investigator, may interfere with participation in the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 subjects were randomized
Pre-assignment Details: Fifteen subjects were randomized to 1 of 4 treatment sequences (ABCD, BACD, ABDC, BADC) in a 1:1:1:1 ratio.
Groups:
- Sequence ABCD: Day 1 (Treatment A): 10 mg dose of RDEA3170, administered as 4 × 2.5 mg ER tablets, in the fasted state; Day 5 (Treatment B): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fasted state; Day 9 (Treatment C): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (low-fat, high-calorie meal); Day 13 (Treatment D): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (high-fat, high-calorie meal).
- Sequence BACD: Day 1 (Treatment B): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fasted state; Day 5 (Treatment A): 10 mg dose of RDEA3170, administered as 4 × 2.5 mg ER tablets, in the fasted state; Day 9 (Treatment C): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (low-fat, high-calorie meal); Day 13 (Treatment D): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (high-fat, high-calorie meal).
- Sequence ABDC: Day 1 (Treatment A): 10 mg dose of RDEA3170, administered as 4 × 2.5 mg ER tablets, in the fasted state; Day 5 (Treatment B): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fasted state; Day 9 (Treatment D): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (high-fat, high-calorie meal); Day 13 (Treatment C): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (low-fat, high-calorie meal).
- Sequence BADC: Day 1 (Treatment B): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fasted state; Day 5 (Treatment A): 10 mg dose of RDEA3170, administered as 4 × 2.5 mg ER tablets, in the fasted state; Day 9 (Treatment D): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (high-fat, high-calorie meal); Day 13 (Treatment C): 10 mg dose of RDEA3170, administered as a single 10 mg ER tablet, in the fed state (low-fat, high-calorie meal).
Period: Overall Study
Arm/Group | Sequence ABCD | Sequence BACD | Sequence ABDC | Sequence BADC
Started | 3 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence ABCD: 2.5 mg x 4 tablets qd fasted, 10 mg tablet qd fasted, 10 mg tablet qd fed low-fat, 10 mg tablet qd fed high-fat.
- Total: Total of all reporting groups
Arm/Group | Sequence ABCD | Sequence BACD | Sequence ABDC | Sequence BADC | Total
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (9.8) | 39 (9.7) | 40 (12.3) | 42 (16.0) | 42 (11.9)
Age, Customized [Number; unit: Participants]
  <65 | 3 | 4 | 4 | 4 | 15
  >=65 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 4 | 4 | 4 | 15
Region of Enrollment [Number; unit: Participants]
  United States | 3 | 4 | 4 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of RDEA3170 in fasted condition.
Time Frame: Days 1 and 5 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Treatment A: 10 mg dose of RDEA3170, administered as 4 × 2.5 mg tablets, in the fasted state.
- Treatment B: 10 mg dose of RDEA3170, administered as a single 10 mg tablet, in the fasted state.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 15 | 15
ng/mL | 14.1 [11.7 to 16.8] | 14.9 [11.9 to 18.8]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The sample size is not based on formal power calculations, as this study is designed only to provide an initial assessment of the Pharmacokinetics (PK), Pharmacodynamics (PD), and safety profile of RDEA3170; Mixed Models Analysis; A mixed effect model on the natural log-transformed PK parameters Cmax, AUClast, and AUC∞ with fixed effect for treatment; Geometric Least Squares Mean Ratio (%) = 107, 90% CI 2-sided [95.2 to 120]

2. Primary Outcome: Time of Occurrence of Maximum Observed Concentration (Tmax)
Description: Tmax of RDEA3170 following various treatments.
Time Frame: Days 1 and 5 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Median (Full Range); unit: hr
Groups:
- Treatment C: 10 mg dose of RDEA3170, administered as a single 10 mg tablet, in the fed state (low-fat, high calorie meal).
- Treatment D: 10 mg dose of RDEA3170, administered as a single 10 mg tablet, in the fed state (high-fat, high calorie meal).
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 15 | 15 | 15 | 15
hr | 2.00 [1.00 to 6.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 6.00] | 4.00 [1.50 to 8.00]

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Quantifiable Last Sampling Timepoint (AUC Last)
Description: AUC last of RDEA3170 in fasted condition.
Time Frame: Days 1 and 5 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 15 | 15
ng·hr/mL | 119 [96.8 to 146] | 114 [85.7 to 153]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The sample size is not based on formal power calculations, as this study is designed only to provide an initial assessment of the PK, PD, and safety profile of RDEA3170; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 97.3, 90% CI 2-sided [85.6 to 111]

4. Primary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC∞)
Description: AUC∞ of RDEA3170 the fasted condition.
Time Frame: Days 1 and 5 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 15 | 15
ng·hr/mL | 131 [105 to 164] | 130 [95.9 to 176]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 100, 90% CI 2-sided [87.3 to 115]

5. Primary Outcome: Apparent Terminal Half-life (t1/2)
Description: t1/2 of RDEA3170 following various treatments.
Time Frame: Days 1 and 5 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 15 | 15 | 15 | 15
hr | 16.5 [11.6 to 23.4] | 15.5 [10.6 to 22.5] | 15.4 [11.6 to 20.4] | 16.6 [11.5 to 23.9]

6. Primary Outcome: Cmax: Effect of High Fat Meal on the PK of RDEA3170 Tablets
Description: Cmax of RDEA3170 in high-fat fed state.
Time Frame: Days 1 to 13 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Treatment B | Treatment D
Number analyzed (Participants) | 15 | 15
ng/mL | 14.9 [11.9 to 18.8] | 27.2 [20.2 to 36.6]
Statistical Analysis 1: Comparison: Treatment B vs Treatment D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 182, 90% CI 2-sided [144 to 230]

7. Primary Outcome: AUC Last: Effect of High Fat Meal on the PK of RDEA3170 Tablets
Description: AUC last of RDEA3170 in high-fat fed state.
Time Frame: Days 1 to 13 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment B | Treatment D
Number analyzed (Participants) | 15 | 15
ng·hr/mL | 114 [85.7 to 153] | 160 [130 to 199]
Statistical Analysis 1: Comparison: Treatment B vs Treatment D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 140, 90% CI 2-sided [121 to 163]

8. Primary Outcome: AUC∞: Effect of High Fat Meal on the PK of RDEA3170 Tablets
Description: AUC∞ of RDEA3170 in high-fat fed state.
Time Frame: Days 1 to 13 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment B | Treatment D
Number analyzed (Participants) | 15 | 15
ng·hr/mL | 130 [95.9 to 176] | 173 [137 to 219]
Statistical Analysis 1: Comparison: Treatment B vs Treatment D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 134, 90% CI 2-sided [114 to 156]

9. Primary Outcome: Cmax: Effect of Low Fat Meal on the PK of RDEA3170 Tablets
Description: Cmax of RDEA3170 in low-fat fed state.
Time Frame: Days 1 to 9 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 15
ng/mL | 14.9 [11.9 to 18.8] | 11.8 [9.23 to 15.1]
Statistical Analysis 1: Comparison: Treatment B vs Treatment C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 79.1, 90% CI 2-sided [66.4 to 94.2]

10. Primary Outcome: AUC Last: Effect of Low Fat Meal on the PK of RDEA3170 Tablets
Description: AUC last of RDEA3170 in low-fat fed state.
Time Frame: Days 1 to 9 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 15
ng·hr/mL | 114 [85.7 to 153] | 97.8 [77.3 to 124]
Statistical Analysis 1: Comparison: Treatment B vs Treatment C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 85.5, 90% CI 2-sided [73.9 to 98.8]

11. Primary Outcome: AUC∞: Effect of Low Fat Meal on the PK of RDEA3170 Tablets
Description: AUC∞ of RDEA3170 in low-fat fed state.
Time Frame: Days 1 to 9 at predose, 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose.
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 15
ng·hr/mL | 130 [95.9 to 176] | 108 [84.4 to 139]
Statistical Analysis 1: Comparison: Treatment B vs Treatment C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio (%) = 83.4, 90% CI 2-sided [73.5 to 94.7]

12. Secondary Outcome: Single Dose Pharmacodynamics (PD) Profile of RDEA3170 From Serum and Urine
Description: PD profiles of uric acid from serum and urine. PD parameters were evaluated to assess whether any potential differences in PK for the 2 different tablets resulted in differences in uric acid excretion.
Time Frame: Day -1: -24, -23, -22, -21, -20, -18, -16, -14, and -12 hours predose. Days 1, 5, 9, and 13: predose (within 30 minutes prior to dosing) and 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 15 | 15 | 15 | 15
Percent
  Serum Urate Maximum % Change | -34.4 (2.08) | -34.4 (2.27) | -37.3 (1.89) | -49.0 (1.96)
  Urine Uric Acid % Change(0-24h) | 96.6 (12.5) | 78.5 (8.38) | 53.4 (8.85) | 65.9 (9.70)
  Renal Clearance of Uric Acid % Change (0-24h) | 170 (19.5) | 147 (15.6) | 128 (18.9) | 179 (21.5)
  Fractional Excretion of Uric Acid % Change (0-24h) | 159 (15.1) | 151 (22.0) | 149 (22.7) | 199 (23.2)

13. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Time Frame: 7 weeks.
Measure: Number; unit: Number of Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 15 | 15 | 15 | 15
Number of Participants | 0 | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: Overall number of baseline participants used to determine number of participants at risk.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 1/15 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=15) | Treatment B (N=15) | Treatment C (N=15) | Treatment D (N=15)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.